CLINICAL TRIAL: NCT06212622
Title: Is the Rate of Early Mobilisation in Hip Fracture Patients Using Alfentanil Better Than Standard Opioid Analgesia (REHAB): a Prospective Cohort Study
Brief Title: Is the Rate of Early Mobilisation in Hip Fracture Patients Using Alfentanil Better Than Standard Opioid Analgesia?
Acronym: REHAB
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC23143
Record Dates: First submitted 2023-12-20; First posted 2024-01-19 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Hip Injuries; Hip Fractures; Pain; Post Operative Pain; Early Ambulation
Keywords: early mobilisation; hip fracture; pain; oxycodone; alfentanil; ambulation
MeSH Terms: conditions — Hip Injuries; Hip Fractures; Pain; Pain, Postoperative | interventions — Alfentanil; Oxycodone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- STANDARD CARE WITH ORAL OXYCODONE: These patients will receive oral oxycodone prior to their post operative day 1 and 2 physiotherapy sessions
  The dose is age dependent (and also on frailty status):
  < 65 years old: Oxycodone 5mg immediate release
  65 - 85 years old: Oxycodone 4mg immediate release
  > 85 years old: Oxycodone 3mg immediate release
  <50kg or particularly frail: Oxycodone 2mg immediate release
  Interventions: Drug: Oxycodone
- INTERVENTION GROUP WITH SUBCUTANEOUS ALFENTANIL: These patients will receive subcutaneous alfentanil prior to their post operative day 1 and 2 physiotherapy sessions
  This is 100 micrograms as a subcutaneous injection
  Interventions: Drug: Alfentanil

INTERVENTIONS:
Drug: Alfentanil — Subcutaneous injection
  Groups: INTERVENTION GROUP WITH SUBCUTANEOUS ALFENTANIL
Drug: Oxycodone — Oral solution
  Groups: STANDARD CARE WITH ORAL OXYCODONE

SUMMARY:
Hip fracture injuries are linked with increased morbidity, frailty, and mortality risk. Studies have shown that in hip fracture surgery, early mobilisation confers better pain control, 30-day complication and mortality rates and could reduce in hospital length of stay.

Though early mobilisation may provide numerous post operative benefits, there are barriers to achieving this reliably and effectively. One such difficulty is pain.

In the Royal Infirmary of Edinburgh (RIE) like many boards across Scotland, oral oxycodone has been routinely used as analgesia to help with post operative pain, in patients who have undergone orthopaedic trauma injuries. However, this analgesic modality is utilised to help with general post operative pain, rather than targeted abolition of pain prior to physiotherapy.

Alfentanil is a relatively new medication which has a very rapid onset of action and short half life. Alfentanil may prove to be a superior form of analgesia for the purpose of encouraging early mobilisation after hip fracture surgery. This study could provide robust evidence for regular use of alfentanil prior to physiotherapy in early post operative hip fracture surgery patients.

DETAILED DESCRIPTION:
Hip fractures are amongst the most common orthopaedic injuries. These fractures predominantly occur in the elderly population, secondary to osteoporosis. Projection studies from across the world suggest that incidence rates of hip fractures are set to increase. Worldwide projections indicate that hip fracture cases will double from 1.26 million in 1990, to 2.6 million by 2025, and to 4.5 million by 2050. The National Joint Registry reports that the number of hip fractures have increased from 1,371 in 2010 to 84,998 in 2021 across England, Wales and Northern Ireland. The Scottish Hip Fracture Audit identifies an increase from 6,369 hip fracture cases in 2007 to 8,380 in 2022. Given the exponential rise in the frail elderly population, these numbers will only further rise in the future.

Hip fracture injuries are linked with increased morbidity, frailty, and mortality risk. Moreover, there is significant social and economic costs on the healthcare system stemming from these injuries. In the United States, these costs are greater than $5.96 billion, annually. In the United Kingdom, these costs are approximately £1.1 billion. Healthcare systems globally, are becoming progressively more financially restrained, and the incidence of hip fractures are set to increase. Thus, further emphasis should be placed on interventions to reduce morbidity and mortality in this frail elderly patient group.

Many studies have shown that early mobilisation after hip fracture surgery provides reduced post operative pain and complication rates and reduces length of stay (LOS) in hospital. Some studies have demonstrated that early ambulation reduces 30-day mortality rates in this patient population. It has been demonstrated that early mobilisation was also associated with an increased rate of discharges directly home, compared to those patients who mobilised late. Although elderly patients have associated co-morbidity and a higher risk of delirium, neither factors influenced inability to mobilise early after surgery. They also found that a greater number of patients who mobilised early were able to be discharged directly home.

Though early mobilisation may provide numerous post operative benefits, there are barriers to achieving this reliably and effectively. One such difficulty is pain. Studies report that pain is often a key obstacle to early ambulation after surgery. In the Royal Infirmary of Edinburgh (RIE) like many boards across Scotland, oral oxycodone has been routinely used as analgesia to help with post operative pain, in patients who have undergone orthopaedic trauma injuries. However, this analgesic modality is utilised to help with general post operative pain, rather than targeted abolition of pain prior to physiotherapy.

Oxycodone has been utilised in clinical practice since 1917. There is in depth literature on the pharmacokinetics of oxycodone. The onset of action of oral oxycodone is between 10-30 minutes. Peak onset occurs around 1 hour. Plasma half-life is 3-5 hours, regardless of route of administration.

On the other hand, alfentanil is relatively new, and the literature is scarce on its pharmacokinetic properties. There is consensus amongst the literature that onset of action of alfentanil is very rapid, with peak onset of intravenous alfentanil as quick as 2 minutes. Plasma half-life of oral alfentanil is 1-2 hours. Moreover, side effects of respiratory depression are lower than that from fentanyl or sufentanil. The combination of rapid onset of pain relief, with an equally quick excretion, makes this medication appealing in palliative care medicine, in which patients are typically frail. This is particularly the case in patients with renal impairment since this medication is excreted by the liver.

Alfentanil may prove to be a superior form of analgesia for the purpose of encouraging early mobilisation after hip fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

* Listed for urgent hip fracture surgery - dynamic hip screw/cannulated hip screw/hemiarthroplasty/total hip arthroplasty/intramedullary nail
* Sustained an insufficiency/low energy type hip fracture
* Male or female aged over 60
* Able to provide informed consent

Exclusion Criteria:

* Pathological or periprosthetic hip fracture
* Mechanism of injury for hip fracture was of high energy
* Patient is unable to comply with the study protocol or functional assessments
* Patients aged less than 60
* Patients who were wheelchair bound prior to injury
* Inability to understand the patient information for the study, provide written informed consent or answer study questionnaires for cognitive or language reasons
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Enrolment in existing research studies

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants listed for urgent hip fracture surgery, after sustaining a hip fracture surgery under the care of participating surgeons at the institution of RIE. 64 participants will be included in this prospective cohort study, 32 in each cohort. There will be consecutively recruitment and follow all hip fracture patients admitted over a month at RIE.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale score | On post operative day 1
  Pain assessment using the visual analogue scale. This is a visual scale measured from 0 to 10, where 0 is no pain and 10 is very severe pain.
Ability to mobilise | On post operative day 1
  Ability to mobilise based on pre assigned physiotherapy levels (PT):
  * PT level 1 -> standing transfer: ability to weight bear on both legs, and transferring from bed to chair without stepping. Equipment will be utilised to help the patient swing round from bed to chair (sara steady/sam hall turner)
  * PT level 2 -> stepping transfer: ability to weight bear on both legs, and transferring from bed to chair with stepping. Equipment will be utilised to help support the patient when stepping (gutter frame/Zimmer frame)
  * PT level 3A -> mobilising to the toilet with assistance of two people
  * PT level 3B -> mobilising to the toilet with assistance of one person
  * PT level 3C -> mobilising to the toilet without assistance

SECONDARY OUTCOMES:
Visual analogue scale score | On post operative day 2
  Pain assessment using the visual analogue scale. This is a visual scale measured from 0 to 10, where 0 is no pain and 10 is very severe pain.
Ability to mobilise | On post operative day 2
  Ability to mobilise based on pre assigned physiotherapy levels (PT):
  * PT level 1 -> standing transfer: ability to weight bear on both legs, and transferring from bed to chair without stepping. Equipment will be utilised to help the patient swing round from bed to chair (sara steady/sam hall turner)
  * PT level 2 -> stepping transfer: ability to weight bear on both legs, and transferring from bed to chair with stepping. Equipment will be utilised to help support the patient when stepping (gutter frame/Zimmer frame)
  * PT level 3A -> mobilising to the toilet with assistance of two people
  * PT level 3B -> mobilising to the toilet with assistance of one person
  * PT level 3C -> mobilising to the toilet without assistance
EuroQol five dimension (EQ-5D) - 5L patient reported outcome measure | At post operative day (POD) 1, POD2, POD 7 and POD 30
  The EQ-5D-5L consists of questions in domains of mobility, self-care, usual activities of daily living, pain/discomfort and anxiety/depression. There are five options for marking severity for each domain. There is also a VAS, rating how the patient perceives health related quality of life from 0-100.
In hospital length of stay | From date of admission until the date of discharge from hospital or date of death, whichever came first (assessed up to 52 weeks)
  In hospital length of stay will be calculated as the number of days in hospital, from the date of admission to the day of discharge.
Total use of analgesia over post operative day 1 and post operative day 2 | post operative day 1 and post operative day 2
  This outcome will be assessed to determine if early mobilisation helps reduce overall postoperative pain during in hospital admission, and see if differing analgesic modalities has any effect on this.
Complication rates and 30-day mortality | At post operative day (POD) 1, POD2, POD 7 and POD 30
  Each patient will be followed up, via their internal TRAKcare patient notes to determine 30-day mortality. Complication rates will be assessed at POD 1, POD 2 and POD 7 alongside the EQ-5D-5L questionnaire. They will also then be followed up at 30 days to assess any further complications. The following complications will be assessed:
  * Any complication
  * Post operative delirium
  * Surgical site infection
  * Wound dehiscence
  * Pneumonia
  * Pulmonary embolism
  * Acute kidney injury
  * Urinary tract infection
  * Cerebrovascular accident
  * Cardiac arrest
  * Myocardial infarction
  * Deep vein thrombosis
  * Delirium
  * Sepsis
  * Mortality
  * Dislocation
  * Re-operation (and reason for this)
  * Readmission (and reason(s) for this)
Discharge destination | Pre admission location will be assessed on the date of admission. Discharge destination will be sought, on the date of discharge from hospital (assessed up to 52 weeks)
  The discharge destination will be sought, and compared with pre-admission status (e.g. at home/care home/residual home), to determine if analgesic modality affects discharge destination

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Clement, MBBS, MD, PhD, FRCS (T&O), Principal Investigator — NHS Lothian
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cummings SR, Black DM, Nevitt MC, Browner W, Cauley J, Ensrud K, Genant HK, Palermo L, Scott J, Vogt TM. Bone density at various sites for prediction of hip fractures. The Study of Osteoporotic Fractures Research Group. Lancet. 1993 Jan 9;341(8837):72-5. doi: 10.1016/0140-6736(93)92555-8. PMID 8093403
- [Background] Kazley J, Bagchi K. Femoral Neck Fractures. StatPearls [Internet]. 2023 May 8 [cited 2023 Sep 1]; Available from: https://www.ncbi.nlm.nih.gov/books/NBK537347/
- [Background] Brittain R, Howard P, Lawrence S, Stonadge J, Wilkinson M, Wilton T, et al. NJR statistical analysis, support and associated services National Joint Registry | 19th Annual Report. [cited 2023 Sep 1]; Available from: www.njrcentre.org.uk
- [Background] Health Scotland P. Scottish Hip Fracture Audit Report 2023 Reporting on episodes of hip fractures in 2022 A Management Information release for Scotland
- [Background] Scottish Hip Fracture Audit Report 2008 Contents. 2006 [cited 2023 Sep 1]; Available from: www.shfa.scot.nhs.uk
- [Background] Kingston A, Comas-Herrera A, Jagger C; MODEM project. Forecasting the care needs of the older population in England over the next 20 years: estimates from the Population Ageing and Care Simulation (PACSim) modelling study. Lancet Public Health. 2018 Sep;3(9):e447-e455. doi: 10.1016/S2468-2667(18)30118-X. Epub 2018 Aug 31. PMID 30174210
- [Background] Downey C, Kelly M, Quinlan JF. Changing trends in the mortality rate at 1-year post hip fracture - a systematic review. World J Orthop. 2019 Mar 18;10(3):166-175. doi: 10.5312/wjo.v10.i3.166. eCollection 2019 Mar 18. PMID 30918799
- [Background] Gdalevich M, Cohen D, Yosef D, Tauber C. Morbidity and mortality after hip fracture: the impact of operative delay. Arch Orthop Trauma Surg. 2004 Jun;124(5):334-40. doi: 10.1007/s00402-004-0662-9. Epub 2004 Apr 17. PMID 15095097
- [Background] Schnell S, Friedman SM, Mendelson DA, Bingham KW, Kates SL. The 1-year mortality of patients treated in a hip fracture program for elders. Geriatr Orthop Surg Rehabil. 2010 Sep;1(1):6-14. doi: 10.1177/2151458510378105. PMID 23569656
- [Background] Adeyemi A, Delhougne G. Incidence and Economic Burden of Intertrochanteric Fracture: A Medicare Claims Database Analysis. JB JS Open Access. 2019 Feb 27;4(1):e0045. doi: 10.2106/JBJS.OA.18.00045. eCollection 2019 Mar 27. PMID 31161153
- [Background] Christodoulou C, Cooper C. What is osteoporosis? Postgrad Med J. 2003 Mar;79(929):133-8. doi: 10.1136/pmj.79.929.133. PMID 12697910
- [Background] Johnell O. The socioeconomic burden of fractures: today and in the 21st century. Am J Med. 1997 Aug 18;103(2A):20S-25S; discussion 25S-26S. doi: 10.1016/s0002-9343(97)90023-1. PMID 9302894
- [Background] Leal J, Gray AM, Prieto-Alhambra D, Arden NK, Cooper C, Javaid MK, Judge A; REFReSH study group. Impact of hip fracture on hospital care costs: a population-based study. Osteoporos Int. 2016 Feb;27(2):549-58. doi: 10.1007/s00198-015-3277-9. Epub 2015 Aug 19. PMID 26286626
- [Background] Heiden JJ, Goodin SR, Mormino MA, Siebler JC, Putnam SM, Lyden ER, Tao MA. Early Ambulation After Hip Fracture Surgery Is Associated With Decreased 30-Day Mortality. J Am Acad Orthop Surg. 2021 Mar 1;29(5):e238-e242. doi: 10.5435/JAAOS-D-20-00554. PMID 32694326
- [Background] Kuru T, Olcar HA. Effects of early mobilization and weight bearing on postoperative walking ability and pain in geriatric patients operated due to hip fracture: a retrospective analysis. Turk J Med Sci. 2020 Feb 13;50(1):117-125. doi: 10.3906/sag-1906-57. PMID 31742370
- [Background] Tan S, Vasireddy A. Early mobilisation following fragility hip fracture surgery: current trends and association with discharge outcomes in a local tertiary hospital. Singapore Med J. 2023 Dec;64(12):721-727. doi: 10.11622/smedj.2021132. PMID 34617696
- [Background] Warren J, Sundaram K, Anis H, McLaughlin J, Patterson B, Higuera CA, Piuzzi NS. The association between weight-bearing status and early complications in hip fractures. Eur J Orthop Surg Traumatol. 2019 Oct;29(7):1419-1427. doi: 10.1007/s00590-019-02453-z. Epub 2019 May 27. PMID 31134326
- [Background] Ferris H, Brent L, Coughlan T. Early mobilisation reduces the risk of in-hospital mortality following hip fracture. Eur Geriatr Med. 2020 Aug;11(4):527-533. doi: 10.1007/s41999-020-00317-y. Epub 2020 Apr 9. PMID 32297275
- [Background] Baer M, Neuhaus V, Pape HC, Ciritsis B. Influence of mobilization and weight bearing on in-hospital outcome in geriatric patients with hip fractures. SICOT J. 2019;5:4. doi: 10.1051/sicotj/2019005. Epub 2019 Feb 28. PMID 30816088
- [Background] Goubar A, Martin FC, Potter C, Jones GD, Sackley C, Ayis S, Sheehan KJ. The 30-day survival and recovery after hip fracture by timing of mobilization and dementia : a UK database study. Bone Joint J. 2021 Jul;103-B(7):1317-1324. doi: 10.1302/0301-620X.103B7.BJJ-2020-2349.R1. PMID 34192935
- [Background] Oldmeadow LB, Edwards ER, Kimmel LA, Kipen E, Robertson VJ, Bailey MJ. No rest for the wounded: early ambulation after hip surgery accelerates recovery. ANZ J Surg. 2006 Jul;76(7):607-11. doi: 10.1111/j.1445-2197.2006.03786.x. PMID 16813627
- [Background] Barone A, Giusti A, Pizzonia M, Razzano M, Oliveri M, Palummeri E, Pioli G. Factors associated with an immediate weight-bearing and early ambulation program for older adults after hip fracture repair. Arch Phys Med Rehabil. 2009 Sep;90(9):1495-8. doi: 10.1016/j.apmr.2009.03.013. PMID 19735776
- [Background] Robinson KP, Wagstaff KJ, Sanghera S, Kerry RM. Postoperative pain following primary lower limb arthroplasty and enhanced recovery pathway. Ann R Coll Surg Engl. 2014 May;96(4):302-6. doi: 10.1308/003588414X13946184900525. PMID 24780024
- [Background] Ramsay MA. Acute postoperative pain management. Proc (Bayl Univ Med Cent). 2000 Jul;13(3):244-7. doi: 10.1080/08998280.2000.11927683. No abstract available. PMID 16389390
- [Background] Kalso E. Oxycodone. J Pain Symptom Manage. 2005 May;29(5 Suppl):S47-56. doi: 10.1016/j.jpainsymman.2005.01.010. PMID 15907646
- [Background] Sadiq NM, Dice TJ, Mead T. Oxycodone. 2024 Feb 20. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482226/ PMID 29489158
- [Background] Lugo RA, Kern SE. The pharmacokinetics of oxycodone. J Pain Palliat Care Pharmacother. 2004;18(4):17-30. doi: 10.1300/j354v18n04_03. PMID 15760805
- [Background] Olesen AE, Upton R, Foster DJ, Staahl C, Christrup LL, Arendt-Nielsen L, Drewes AM. A pharmacokinetic and pharmacodynamic study of oral oxycodone in a human experimental pain model of hyperalgesia. Clin Pharmacokinet. 2010 Dec;49(12):817-27. doi: 10.2165/11536610-000000000-00000. PMID 20873879
- [Background] Poyhia R, Seppala T, Olkkola KT, Kalso E. The pharmacokinetics and metabolism of oxycodone after intramuscular and oral administration to healthy subjects. Br J Clin Pharmacol. 1992 Jun;33(6):617-21. doi: 10.1111/j.1365-2125.1992.tb04090.x. PMID 1389934
- [Background] Ordonez Gallego A, Gonzalez Baron M, Espinosa Arranz E. Oxycodone: a pharmacological and clinical review. Clin Transl Oncol. 2007 May;9(5):298-307. doi: 10.1007/s12094-007-0057-9. PMID 17525040
- [Background] Ferraz Goncalves JA, Sousa F, Alves L, Liu P, Coelho S. Use of Alfentanil in Palliative Care. Pharmacy (Basel). 2020 Dec 16;8(4):240. doi: 10.3390/pharmacy8040240. PMID 33339325
- [Background] Moman RN, Mowery ML, Kelley B. Alfentanil. 2024 Jan 11. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK470456/ PMID 29261876